CLINICAL TRIAL: NCT00582257
Title: Early Onset and Familial Gastric Cancer Registry
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); Queens Health Network (Other); University of Southern California (Other); Shaare Zedek Medical Center (Other); Obafemi Awolowo University Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 05-118
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Stomach Cancer; 05-118
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surveys and Questionnaires; Masks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Germline DNA and Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High Genetic Risk:: Early Onset Gastric Cancer - diagnosis of gastric cancer before the age of 50 without a family history of the disease.
  Familial Gastric Cancer - having a family history of gastric cancer as defined as one first degree relative or 2 second degree relatives.
  Relative - Relatives of participants eligible for the High Genetic Risk Cohort will be eligible for participation. These relatives may also be at high risk of developing gastric cancer. These individuals will fall under the Cancer Cohort. Eligible relatives will be defined as someone having a relative who meets criteria for either the Early Onset Cancer Cohort or the Familial Gastric Cancer Cohort, or having a family history of a genetic mutation known to be associated with gastric cancer.
  Interventions: Behavioral: questionnaires
- Low Genetic Risk: Closed to Accrual: Sporadic Gastric Cancer - gastric cancer that appears to have occurred by random or sporadic mutation. Specifically, a patient with gastric cancer not eligible for either High Genetic Risk cohort.
  Control (closed to accrual) - A participant that is not a blood relative of a patient or relative participant, without gastric cancer and without a family history of a CDH1 gene mutation. Select MSK participants with Hereditary Diffuse Gastric Cancer with identified CDH1 germline genetic mutation will be invited by MSKCC only to complete the onetime Pre-implantation Genetic Diagnosis (HDGC PGD) survey. These patients may be verbally consented over the telephone.
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Participation in the registry will consist of adequately completing the family history questionnaire (one per family) the gastric cancer risk factor questionnaire and providing a blood sample for future correlative studies. Registry participants (both Patient/Relative and Control cohorts) will be required to submit tissue (both normal and/or tumor) to create a Tissue and DNA repository. Select participants will be invited to undergo Genetic Counseling, eg. those participants who meet clinical criteria for HDGC.
  Other Names: At outside centers, recruitment procedures are similar to the procedures at; MSK with the following two exceptions: Due to practice patterns, it may not; be feasible to obtain "Control Cohort" patients. Collaborating sites may; participate in the study without opening a "Control Cohort" after discussion; with the study PI. Phone consenting will only be done at MSKCC.

SUMMARY:
The purpose of this study is to establish a gastric cancer registry. A registry is a database of information. With the registry, we can learn more about the genetic causes of gastric cancer in order to develop better methods of early diagnosis, prevention, and treatment of gastric cancers. As part of this study, you will be asked to join a registry of families who are affected with various forms of gastric cancer. These registries are important because they may help physicians better manage gastric cancer now and in the future. Participating in the Early Onset and Familial Gastric Cancer Registry can also be educational for families, since it will provide important information to patients, families, and physicians. All of this will help to further our understanding of genetic causes of gastric cancer and eventually, help determine better ways to diagnose, treat, and survey patients with gastric cancer and people who may have a higher risk for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Patient/Relative Cohort:

Must meet one or more criteria below:

1. A person with a diagnosis of gastric or gastroesophageal junction (GEJ) adenocarcinoma confirmed at the treating institution.
2. A person without gastric or GEJ adenocarcinoma who has or had a first degree relative eligible for a High Risk Genetic sub-group (EOGC/FGC).

   1. Early Onset Gastric Cancer - diagnosis of gastric cancer before the age of 50 without a family history of the disease.
   2. Familial Gastric Cancer - having a family history of gastric cancer as defined as one first degree relative or 2 second degree relatives.
3. A person without gastric or GEJ adenocarcinoma who has a personal family history of a genetic mutation associated with the development of gastric or GEJ adenocarcinoma (i.e. family history of CDH1 mutation).

II. Must be willing to provide a blood sample for germline DNA. These individuals will sign the "Patient/Relative Consent". Following enrollment, we will assign individuals to the appropriate High Genetic Risk or Low Genetic Risk groups based on the age of diagnosis and their family history.

Subject Exclusion Criteria

Patients are ineligible for the study if they:

* Have any condition, which in the opinion of the primary MSK clinician or investigators precludes their ability to provide informed consent.
* Relatives of patients that are not eligible for the High Genetic Risk Cohorts who are less than 18 years of age are excluded.
* Relatives of patients eligible for the High Genetic Risk Cohorts who do not have a proband available to join the study are excluded. (Unless there is a known CDH1 mutation in the family).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at MSK or collaborating centers. If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participation and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study.
Sampling Method: Non-Probability Sample
Enrollment: 971 (Actual)
Dates: Start 2005-12-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Create registry of families w/ early onset & familial gastric cancer for analysis of risk factors, family history and unidentified susceptibility genes. Create cohorts of pts w/ low genetic risk for the development of gastric cancer | December 2010

SECONDARY OUTCOMES:
To determine the incidence of CDH1 germline mutations among individuals with early onset or familial gastric cancer and their relatives. | December 2010
To determine the gastric pathology evident from a single baseline endoscopic screen of unaffected first-degree relatives of a patient with EOGC or FGC. | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: David Kelsen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (9):
  - University of Southern California - Norris Cancer Hospital, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
- Obafemi Awolowo University Teaching Hospital, Ile-Ife, Nigeria

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center website — http://www.mskcc.org